CLINICAL TRIAL: NCT01699113
Title: Effects of YF476, a Gastrin Antagonist, and Rabeprazole, a Proton Pump Inhibitor, Alone and in Combination, on Gastric Function in Healthy Subjects
Brief Title: Effects of YF476 and Rabeprazole on Gastric Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trio Medicines Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 05-021
Record Dates: First submitted 2012-09-26; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Hypergastrinaemia
Keywords: YF476; gastrin receptor antagonist; gastric pH; gastrin; rabeprazole; proton-pump inhibitor; gastric function; healthy subjects
MeSH Terms: interventions — YF 476; Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: YF476 — Subjects will be randomised to once daily treatment by mouth for 6 weeks with:
  * YF476 100 mg; or
  * rabeprazole 20 mg; or
  * a combination of YF476 100 mg and rabeprazole 20 mg.
Drug: Rabeprazole — Subjects will be randomised to once daily treatment by mouth for 6 weeks with:
  * YF476 100 mg; or
  * rabeprazole 20 mg; or
  * a combination of YF476 100 mg and rabeprazole 20 mg.

SUMMARY:
The primary objectives are to find out in healthy subjects if:

* YF476 prevents the ECL-cell hyperplasia induced by repeated doses of rabeprazole - a proton pump inhibitor;
* YF476 also prevents rebound hyperacidity after stopping rabeprazole; and
* YF476 by itself causes neither ECL-cell hyperplasia after repeated doses nor rebound hyperacidity after stopping YF476.

The secondary objectives are to:

* assess the safety and tolerability of YF476, alone and in combination with rabeprazole;
* compare the effects of YF476, alone and in combination with rabeprazole, on serum gastrin and plasma CgA and SST;
* assess if there is a pharmacokinetic interaction between YF476 and rabeprazole;
* assess the pharmacokinetics of repeat doses of YF476 by itself; and
* study the metabolism of YF476.

DETAILED DESCRIPTION:
We want to know if YF476 prevents ECL-cell hyperplasia induced by PPI, and rebound hyperacidity after PPI withdrawal, in man, as it does in the rat. A positive result would support further studies to assess if a combination of YF476 and a PPI is a better way of treating patients with peptic ulcer disease and GORD than a PPI alone. Equally, we want to know if YF476 by itself not only inhibits gastric acid secretion but also does not cause ECL-cell hyperplasia and rebound hyperacidity after withdrawal. A positive result would support further studies to assess if YF476 alone is an alternative and perhaps better treatment for patients with peptic ulcer disease and GORD than a PPI alone. The study design is important. We need to ask ourselves several questions.

First, which PPI should we use? Omeprazole has been studied more than other PPI, and is probably still the most widely used PPI in the clinic. A disadvantage of omeprazole is that its metabolism is affected by genetic polymorphism. Studies of human liver microsomes in vitro (Yamazaki et al 1997) show that omeprazole is metabolised by 5-hydroxylation (catalysed by CYP2C19, and to a lesser extent CYP3A4) and sulphoxidation (catalysed by CYP3A4). YF476 inhibits CYP3A4/5 in vitro; but we don't know how relevant that is in vivo. CYP2C19 has 3 genotypes: homozygous extensive metabolisers, with higher enzymatic activity; heterozygous extensive metabolisers, with moderate enzymatic activity; and poor metabolisers, with markedly impaired enzymatic activity. Consequently, in CYP2C19 homozygous extensive metabolisers, acid suppression by omeprazole is reduced compared with heterozygous and poor metabolisers (Shirai et al 2001). Homozygous extensive metabolisers comprise about 70% of the European and USA populations and about 30% of the Asian population. Recently, a new CYP2C19 gene variant that causes ultrarapid metabolism of omeprazole has been identified in 18% of Swedes (Sim et al 2006). So, if we use omeprazole, we should genotype subjects for CYP2C19. Ideally, we should stratify their allocation to treatments, to try to avoid confounding the results. But, we are unlikely to be able to get the genotyping results quickly enough after screening to make stratification practical.

Rabeprazole, unlike omeprazole, is metabolised mainly via a non-enzymatic pathway with minor CYP2C19 and CYP3A4 involvement. Therefore, acid suppression by rabeprazole is less affected by CYP2C19 genotype (Shirai et al 2001; Miura et al 2006), which is one reason for using rabeprazole instead of omeprazole. Omeprazole and rabeprazole are both off-patent, so a combination product of YF476 and either PPI is possible.

Second, what dose of PPI should we use, and for how long? The dose of PPI should be one that is clinically relevant. If the choice of PPI is omeprazole, the dose should be 40 mg daily, because 20 mg -- the standard clinical dose -- was less effective than the recommended doses of other PPI in raising gastric pH (Warrington et al 2006). Rabeprazole 20 mg was more effective than esomeprazole 20 mg in those studies, another reason for using rabeprazole (Warrington et al 2005). Taking everything into account, we have decided to use rabeprazole 20 mg daily for our study.

The duration of PPI dosing is probably more important than the choice of PPI and dose. The longer the duration of dosing, the more likely we are to show the morphological changes of ECL-cell hyperplasia. But ethical considerations and compliance issues mean that we have to compromise over duration of dosing. The available evidence suggests that 2 weeks is not long enough to induce ECL-cell hyperplasia, whereas 8-12 weeks may be more than long enough. So, 6 weeks seems a reasonable compromise.

Third, how long after stopping the PPI should we assess rebound hyperacidity? Early studies in man failed to show rebound hyperacidity after stopping omeprazole because the assessments were done too soon (Prewett et al 1991). PPIs are non-competitive inhibitors of the proton pump, which takes days to regenerate fully. The available evidence suggests that 2 weeks after PPI withdrawal is long enough to study rebound hyperacidity.

Fourth, what dose of YF476 should we use? Single and repeated doses of 100 mg daily were well tolerated and completely suppressed pentagastrin-stimulated increases in gastric acid volume and H+ content in healthy subjects. The toxicology and toxicokinetic studies support dosing of 100 mg daily for up to 13 weeks. So, a dosing schedule of 100 mg daily for 6 weeks is appropriate.

Fifth, is it safe to give a PPI and YF476 together? No safety problems were reported when rats were given omeprazole and YM022, an enantiomer of YF476, for 13 weeks (Nishida et al 1995). Also, no safety problems were reported when omeprazole and YF476 were given to rats for 8 weeks (Chen et al 2000). However, whatever PPI we use, we should assay blood concentrations of PPI and YF476 (Redrup et al 2002) at the start and end of dosing, lest a drug-drug interaction confound the results of the outcome measures.

Sixth, what tests of gastric function and ECL cells should we use to compare the treatments? We should study: plasma gastrin, to assess the degree of hypergastrinaemia; plasma CgA, a marker of ECL-cell hyperplasia; plasma SST, a marker of D-cell activity; pentagastrin-stimulated increases in gastric acid volume and H+ content, and 24-hour ambulatory pH, to compare anti-secretory responses during and after stopping treatments; gastric biopsies, to assess changes in ECL-cell histology and enzymes; and dyspepsia symptoms, to assess occurrence of symptomatic rebound hyperacidity after stopping treatment.

Seventh, should the study be crossover or parallel-group in design? In healthy subjects, a crossover study is often the ideal design. Comparisons are made within rather than between subjects, which reduces the variability of the results. But, a crossover design is not practical given the long dosage period and the demanding procedures. By using rabeprazole, we avoid the potential problem of between-subject differences attributable to CYP2C19 genetic polymorphism. So, a parallel-group design with 3 groups of subjects randomised to either YF476, rabeprazole, or a combination of YF476 and rabeprazole, is a sensible solution.

Eighth, should we have identical treatments and a placebo group? We can over-encapsulate the treatments to make them identical so that the study is double blind in design. Ideally, we should have a placebo group, but if the study is double blind in design and the methods are mostly objective, a placebo group is not essential.

Finally, should we use patients or healthy subjects? Healthy subjects and patients with peptic ulcer disease or GORD all develop hypergastrinaemia and ECL-cell hyperplasia after repeated dosing with a PPI, and rebound hyperacidity after stopping the PPI. Nevertheless, the study is best done in healthy subjects because they are more likely to comply with the demanding study procedures, more homogeneous, more robust, and not on medication. The YF476 reproductive toxicology studies justify including women who are not at risk of pregnancy. However, H pylori-positive subjects should be excluded. In a recent UK community study, 15% of people were H pylori-positive (Lane et al 2006).

ELIGIBILITY:
Inclusion Criteria:

* Men or women, deemed healthy on the basis of a clinical history, physical examination, ECG and safety tests of blood and urine;
* able to give fully-informed, written consent.

Exclusion Criteria:

* Women who are pregnant, lactating or using a steroid contraceptive.
* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the subject.
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the subject's participation in the trial or make it unnecessarily hazardous.
* Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness.
* Evidence of high serum gastrin at screening or achlorhydria at baseline.
* Presence or history of severe adverse reaction to any drug.
* Use of a prescription medicine or antacids during the 28 days before the trial or use of an over-the-counter medication, with the exception of paracetamol, during the 7 days before the trial.
* Participation in a trial of a new drug substance or a prescription medicine within the previous 3 months.
* Presence or history of drug or alcohol abuse, or intake of more than 28 units of alcohol weekly (for men) or 21 units of alcohol weekly (for women).
* Blood pressure and heart rate in supine position at the screening examination outside the ranges 90-160 mm Hg systolic, 40-95 mm Hg diastolic; heart rate 40_100 beats/min.
* Possibility of the subject not co-operating with requirements of the protocol.
* Evidence of drug abuse on urine testing.
* Positive test for hepatitis B, hepatitis C, HIV1 or HIV2.
* Loss of > 400 mL blood, e.g. blood donation, in the 3 months before the trial.
* Objection by the General Practitioner (GP) to the subject entering the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Measurement of pentagastrin-stimulated gastric volume
Measurement of pentagastrin-stimulated H+ content (titratable acidity)
Measurement of pentagastrin-stimulated pH
Measurement of pentagastrin-stimulated bicarbonate
Histology of ECL cells
  4 biopsy specimens were taken from the oxyntic mucosa of the body of the stomach. The specimens were prepared and coded for blinded analysis.
  The biopsy specimens were analysed by histology, immunohistochemistry of HDC and CgA, and electron microscopy.
Immunostaining of HDC and CgA
  4 biopsy specimens were taken from the oxyntic mucosa of the body of the stomach. The specimens were prepared and coded for blinded analysis.
  The biopsy specimens were analysed by histology, immunohistochemistry of HDC and CgA, and electron microscopy.
Electron microscopy of gastric mucosal biopsies
  4 biopsy specimens were taken from the oxyntic mucosa of the body of the stomach. The specimens were prepared and coded for blinded analysis.
  The biopsy specimens were analysed by histology, immunohistochemistry of HDC and CgA, and electron microscopy.

SECONDARY OUTCOMES:
Measurement of 24-h intragastric pH
Measurement of 24-h serum gastrin
Measurement of 24-h plasma SST and CgA
Measurement of dyspepsia symptoms; antacid usage
Measurement of pharmacokinetics of YF476 in blood and urine
  Blood samples for assay of YF476 and/or rabeprazole: before and frequently up to 24 h after the first dose, and at the end of treatment (Day 40); and before dosing on clinic visits during the treatment period, to assess compliance. 3 additional blood samples (4 mL) on Day 40 for future analysis of metabolites. Urine collection 0-24 h after the first dose and at the end of treatment (Day 40), for future analysis of metabolites.
Measurement of pharmacokinetics of rabeprazole in blood and urine
  Blood samples for assay of YF476 and/or rabeprazole: before and frequently up to 24 h after the first dose, and at the end of treatment (Day 40); and before dosing on clinic visits during the treatment period, to assess compliance. 3 additional blood samples (4 mL) on Day 40 for future analysis of metabolites. Urine collection 0-24 h after the first dose and at the end of treatment (Day 40), for future analysis of metabolites.
Measurement of safety assessments
  Physical examination; vital signs; ECG (especially QTc interval); safety tests of blood and urine
Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Boyce, Study Director — Trio Medicines Limited
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom